CLINICAL TRIAL: NCT00178685
Title: Self-determination and Maintaining Tobacco Abstinence
Brief Title: Smokers' Health Project: Self-Determination and Maintaining Tobacco Abstinence
Acronym: SHP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Rochester (Other)
Collaborators: National Cancer Institute (NCI) (NIH); New York State Department of Health (Other Government); Greater Rochester Area Tobacco Cessation Center (Unknown); Health Maintenance Consortium (Unknown); National Institutes of Health (NIH) (NIH)
Responsible Party: Geoffrey C Williams, University of Rochester, Smokers' Health Project
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 10085; R01 CA10666; 1R21CA119112-01A2 (NIH)
Record Dates: First submitted 2005-09-13; First posted 2005-09-15 (Estimated); Results first posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2009-07

CONDITIONS: Tobacco Use Disorder
Keywords: Self-determination; motivation; adherence; competence; autonomy; tobacco dependence; Tobacco use and dependence; Behavior change
MeSH Terms: conditions — Tobacco Use Disorder; Tobacco Use

STUDY DESIGN:
Who Masked: Outcomes Assessor

INTERVENTIONS:
Behavioral: Self-determination Intervention for Tobacco Dependence — autonomy supported behavioral intervention for tobacco dependent individuals
  Other Names: Smokers' Health Project

SUMMARY:
These two studies will examine the role of autonomous motivation in maintained adherence. The first study will determine whether smokers are still abstinent from tobacco 32 months after starting in a previous project (Smoker's Health Study). The purpose of the second study is to determine which of three treatments for tobacco dependence provides the greatest amount of protection from relapsing to smoking after quitting. Specifically, the investigators will determine if extending the length of treatment time focusing on relapse prevention and arranging for support from important others prevents relapse compared to community care. Also, the investigators will determine if providing extended treatment time and support from important others plus providing medications to those that don't want to quit prevents long term relapse compared to just extending the length of treatment time and support from others. Additionally, a sub set of the population will be randomized to using hand held palm devices to recover real-time data assessment during the last 10 months of the project.

DETAILED DESCRIPTION:
These two studies will extend our examination of self-determination theory (SDT) based counseling interventions to the issue of maintained abstinence from tobacco use. Two projects are proposed, both of which build on the results of our current trial. The first is a 32-month follow-up of the smoking status of patients in the preceding trial called the Smoker's Health Study (self-determination, smoking, diet, and health). That SDT intervention (4 counselor visits over 6 months) increased cessation at 6 months relative to community care, and was also effective in increasing 12 month prolonged abstinence, and the results have been reported in two manuscripts (Williams, McGregor, Sharp, Levesque, Kouides, Ryan, and Deci, In press; Williams, McGregor, Sharp, Levesque, Kouides, Ryan, and Deci, 2005). The part of this first project that will be conducted as part of this grant will be to complete 32 month follow-up of smokers in the Smoker's Health Study. The second project is a 3-cell clinical trial called the Smoker's Health Project that will examine two extensions of the current intervention, both of which place greater emphasis on use of, and adherence to, cessation medications. The two arms will be compared to community care. Both arms involve two visits with a physician to discuss medications and side effects. In both interventions, counselors will address medication adherence. The two arms differ in that patients not ready to quit in one arm will receive a smoking reduction approach (with medications) in which they first try to reduce their smoking to half and then attempt cessation. In addition, to place greater emphasis on medications and to examine medication adherence as a mediator of maintained cessation.

There will be two major changes in the intervention intended to facilitate long-term maintenance. First, the intervention will extend over 12 months (whereas the current one lasts only 6 months) with meetings during the additional 6 months focusing on maintenance and relapse prevention. Second, at least one family member or best friend of each patient will be encouraged to meet with a counselor to learn how to be more autonomy supportive with the patient around issues related to tobacco. Cessation and maintained abstinence will be examined with logistic regression. The SDT process model of maintained cessation will be tested using structural equation modeling, and cost-effectiveness analyses will be done for the interventions.

ELIGIBILITY:
Inclusion Criteria:

* Smoking 5 or more cigarettes per day.
* 18 years of age or older.
* Speak and read English.
* Eligible regardless of desire to quit smoking

Exclusion Criteria:

* Pregnancy
* History of psychotic illness other than depression
* Life expectancy of less than 24 months
* Dementia, or incompetence for medical decision making

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 837 (Actual)
Dates: Start 2004-08; Primary Completion 2008-08 (Actual); Study Completion 2008-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Geoffrey C Williams, MD, Ph.D., Principal Investigator — University of Rochester
Locations (1):
- Smokers' Health Project, Rochester, New York, United States

REFERENCES:
- [Background] Williams GC, McGregor HA, Sharp D, Levesque C, Kouides RW, Ryan RM, Deci EL. Testing a self-determination theory intervention for motivating tobacco cessation: supporting autonomy and competence in a clinical trial. Health Psychol. 2006 Jan;25(1):91-101. doi: 10.1037/0278-6133.25.1.91. PMID 16448302
- [Background] Williams GC, McGregor H, Sharp D, Kouldes RW, Levesque CS, Ryan RM, Deci EL. A self-determination multiple risk intervention trial to improve smokers' health. J Gen Intern Med. 2006 Dec;21(12):1288-94. doi: 10.1111/j.1525-1497.2006.00621.x. PMID 16995893
- [Background] Williams GC, Minicucci DS, Kouides RW, Levesque CS, Chirkov VI, Ryan RM, Deci EL. Self-determination, smoking, diet and health. Health Educ Res. 2002 Oct;17(5):512-21. doi: 10.1093/her/17.5.512. PMID 12408196
- [Derived] Niemiec CP, Ivarsson A, Weman K, Smit E, Williams GC. Self-determination theory and the smoking cessation process: Daily electronic self-reports can identify the initiation of quit attempts. Patient Educ Couns. 2023 Oct;115:107886. doi: 10.1016/j.pec.2023.107886. Epub 2023 Jul 7. PMID 37567038
- [Derived] Williams GC, Niemiec CP, Patrick H, Ryan RM, Deci EL. Outcomes of the Smoker's Health Project: a pragmatic comparative effectiveness trial of tobacco-dependence interventions based on self-determination theory. Health Educ Res. 2016 Dec;31(6):749-759. doi: 10.1093/her/cyw046. Epub 2016 Oct 22. PMID 27923864
- [Derived] Ternullo SR, Abdolahi A, Williams GC. Study of monotherapy versus combination therapy for tobacco dependence among heavily addicted smokers. J Am Pharm Assoc (2003). 2017 Jan-Feb;57(1):77-81.e1. doi: 10.1016/j.japh.2016.08.011. Epub 2016 Nov 11. PMID 27839954
- [Derived] Pesis-Katz I, Williams GC, Niemiec CP, Fiscella K. Cost-effectiveness of intensive tobacco dependence intervention based on self-determination theory. Am J Manag Care. 2011 Oct 1;17(10):e393-8. PMID 21999719
- [Derived] Williams GC, Patrick H, Niemiec CP, Ryan RM, Deci EL, Lavigne HM. The smoker's health project: a self-determination theory intervention to facilitate maintenance of tobacco abstinence. Contemp Clin Trials. 2011 Jul;32(4):535-43. doi: 10.1016/j.cct.2011.03.002. Epub 2011 Mar 5. PMID 21382516
- [Derived] Williams GC, Niemiec CP, Patrick H, Ryan RM, Deci EL. The importance of supporting autonomy and perceived competence in facilitating long-term tobacco abstinence. Ann Behav Med. 2009 Jun;37(3):315-24. doi: 10.1007/s12160-009-9090-y. Epub 2009 Apr 17. PMID 19373517
- [Derived] Niemiec CP, Ryan RM, Deci EL, Williams GC. Aspiring to physical health: the role of aspirations for physical health in facilitating long-term tobacco abstinence. Patient Educ Couns. 2009 Feb;74(2):250-7. doi: 10.1016/j.pec.2008.08.015. Epub 2008 Oct 5. PMID 18838243
- See also: Related Info — http://www.selfdeterminationtheory.org

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruitment began in August 2004 and completed in September 2008. Subjects were consented in the research office.
Groups:
- Community Care: The CC condition was similar to the translated 6-month SDT and PHS Guideline-based intensive intervention validated in the previous trial and provided for the CC subjects who wanted to make a quit attempt. The clinical endpoint was to guide the subjects to be fully autonomous about stopping smoking, including not stopping if not willing to stop smoking. Once willing to stop, the Tobacco Dependence Counselor (TDC, 4 contacts) worked to provide problem solving and skills training as recommended in the PHS Guideline (Chapter 4) and the prescriber (2 visits) guided the subjects to be fully autonomous about use of effective medications. Those not wanting to stop within 30 days of the first appointment were asked to call back when ready.
- Extended Autonomy Support (EAS: The EAS condition provided the same content as CC, but the intervention was extended: (1) from 6 to12 months; (2) to include 8 contacts (six in first 6 months and two in second 6-months); (3) by encouraging smokers to attend treatment, even if not ready to stop; and (4) by asking the smoker to bring an important other (non-health-care professional) to one 50-minute instructional session about how to support the smoker's autonomy.
- Harm Reduction (HR): The HR condition had the same features as EAS, but offered initiation of a first-line smoking cessation medication if unwilling to stop, but willing to reduce their cigarettes by half. Subjects were informed that there is no evidence to suggest that reducing cigarette use improves health, but that doing so might increase their confidence in stopping.
Period: Overall Study
Arm/Group | Community Care | Extended Autonomy Support (EAS | Harm Reduction (HR)
Started | 172 | 324 | 324
Completed | 61 | 120 | 128
Not Completed | 111 | 204 | 196
Not completed — Death | 3 | 3 | 6
Not completed — Lost to Follow-up | 100 | 187 | 183
Not completed — Withdrawal by Subject | 8 | 14 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Community Care | Extended Autonomy Support (EAS | Harm Reduction (HR) | Total
Number analyzed (Participants) | 172 | 324 | 324 | 820
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 163 | 309 | 303 | 775
  >=65 years | 9 | 15 | 21 | 45
Age Continuous [Mean (Standard Deviation); unit: years] | 47.74 (11.49614) | 46.27 (12.14891) | 48.32 (11.69470) | 47.39 (11.69)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 98 | 194 | 196 | 488
  Male | 74 | 130 | 128 | 332

OUTCOME MEASURES:

1. Primary Outcome: 12 Month Prolonged Abstinence From Tobacco Measured at 12 Months From Completion of Intervention.
Description: The primary outcome measure was 12-month prolonged abstinence (12M-PA) assessed by patient self-report 12-months after the intervention ended. If participant responded that they had not smoked a cigarette, even a puff, in the last 7 days at 12 months post-intervention, and reported date of last cigarette was 365 days or more prior to assessment date, then they were considered to have 12 month prolonged abstinence. A baseline-observation-carried-forward (BOCF)strategy was used for missing data such that those not reporting smoking status 12 months post-intervention were considered smoking.
Time Frame: 12 months after subject completes intervention.
Population: A baseline-observation-carried-forward (BOCF)strategy was used for missing data such that those not reporting smoking status 12 months post-intervention were considered smoking.
Measure: Number; unit: participants
Arm/Group | Community Care | Extended Autonomy Support (EAS | Harm Reduction (HR)
Number analyzed (Participants) | 169 | 321 | 318
participants | 169 | 321 | 318

2. Secondary Outcome: 7 Day Point Prevelence (7DPP)
Description: Seven-day point prevalence abstinence (7DPP) was assessed by asking: "Have you smoked a cigarette, even a puff, in the last 7 days?"16 Participants were also asked if they had smoked cigars or pipe, chewed tobacco, or used snuff in the past 7 days, and if they responded yes they were considered tobacco users.
Time Frame: 12 months after the intervention
Population: 820 individuals were randomized to condition, of those, 12 died during the course of the study (all deaths were found to be unrelated to the study). Final analysis number included all those randomized and excluded those who died during the study.
Measure: Number; unit: participants
Arm/Group | Community Care | Extended Autonomy Support (EAS | Harm Reduction (HR)
Number analyzed (Participants) | 169 | 321 | 318
participants | 169 | 321 | 318

ADVERSE EVENTS:
Arm/Group | Community Care | Extended Autonomy Support (EAS | Harm Reduction (HR)
Serious Adverse Events (participants affected / at risk) | 4/172 | 3/324 | 6/324
Other Adverse Events (participants affected / at risk) | 1/172 | 1/324 | 0/324
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community Care (N=172) | Extended Autonomy Support (EAS (N=324) | Harm Reduction (HR) (N=324)
Death (General disorders) | 4 (4) | 3 (3) | 6 (6)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Community Care (N=172) | Extended Autonomy Support (EAS (N=324) | Harm Reduction (HR) (N=324)
Dropped from study after patient quit smoking (Social circumstances) | 1 (1) | 1 (1) | 0 (0) — Unable to locate specific adverse reaction/note from cardiology.Patient dropped from the study 2 weeks after being decreased to 2 -14 mg patches per day & previously had quit smoking.
Patient had adverse event while being treated for MS. Unrelated to smoking study. (General disorders) | 1 (1) | 1 (1) | 0 (0) — Patient was being treated for MS with SoluMedrol. Adverse event unrelated to smoking study.

LIMITATIONS AND CAVEATS:
A limitation of this study is the low completion rate of smokers enrolling in the study. This increases the chance of accepting the null hypothesis when there may be differences between groups if all smokers had provided their outcomes.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No